CLINICAL TRIAL: NCT04764981
Title: Clinical Outcomes of Olfactory Training for Treatment of Olfactory Dysfunction After COVID-19
Brief Title: Olfactory Training for Olfactory Dysfunction After Coronavirus Disease - 19 (COVID-19)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidade do Estado do Pará (Other)
Responsible Party: Principal Investigator, ALNA CAROLINA MENDES PARANHOS, Professor, Universidade do Estado do Pará
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OLFATO001
Record Dates: First submitted 2021-02-14; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Covid19; SARS-CoV Infection; Olfactory Disorder; Anosmia
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Anosmia

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial study, with 2 experimental groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants of groups will be evaluated and random inserted in one of the experimental groups. The person responsible for reassessment will be blinded for which group the individual reassessed came from.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1: Essences Oils (Experimental): The individuals of this group are 150 individuals with olfactory disorder related to COVID-19 that will be submitted to clinical exams, olfactory test and MRI imaging, after that, participants will undergo an olfactory training with essences oils. Each participant in this group will receive a kit with four 30 ml bottles, each containing a circular piece of watercolor paper soaked in one of the four essences oils (rose, eucalyptus, lemon and cloves) used in olfactory training, a manual to make the olfactory training at home and a self-assessment diary which should be filled weekly. Each participant of this group will use the training kit for three months, the olfactory training consists of inhaling each of the substances for 30 seconds, with an interval of 30 seconds between them, twice a day, upon waking up and before bed, the participants will be reassessed with CCCRT after each month of training. The results of this group will be compared with the other groups.
  Interventions: Other: Essence oils
- Experimental Group 2: Clinical follow-up (No Intervention): The individuals of this group are 150 individuals with olfactory disorder related to COVID-19. that will be submitted to clinical exams, olfactory test and MRI imaging, after three months they will be reassessed.
- Control Group (No Intervention): The individuals of this group are 50 healthy individuals, without previous COVID-19 infection, that will be submitted to clinical exams, olfactory test, MRI imaging and the participants will be tested for the ability to identification of the essence oils utilized by Experimental group 1.

INTERVENTIONS:
Other: Essence oils — Consists in olfactory training using essence oils
  Arms: Experimental Group 1: Essences Oils

SUMMARY:
It is a randomized controlled clinical trial study that aims to follow a sample of individuals with persistent olfactory dysfunction post-COVID-19. The aim of this study is assess the clinical outcomes of olfactory training therapy in the treatment of persistent olfactory dysfunctions after COVID-19. The sample will consist of 350 participants, being 300 individuals with persistent olfactory dysfunction post-COVID-19 and 50 healthy individuals. Volunteers' will be separated in two experimental groups (1 and 2 ) and a control group. All participants will be submitted to clinical evaluation that include the Connecticut Chemosensory Clinical Research Test (CCCRT), an olfactory test to diagnose anosmia and hyposmia, and two skull Magnetic Resonance imaging (MRI). Only participants of Experimental group 1 will be submitted to an olfactory training with essences oils. Experimental group 2 will only receive a clinical follow-up after three months and control group will be only submitted to neurological exam, olfactory test, MRI imaging and test their ability to discriminate the essence oils used in olfactory training. As a result, is expected a better understanding of the characteristics of olfactory dysfunction caused by Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) virus infection, as well as the effectiveness and viability of using Olfactory Training as a therapeutic alternative.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COVID-19 by Real Time Polymerase chain-reaction for SARS-CoV-2 or serological tests for SARS-CoV-2 antigens.\
* Olfactory dysfunction confirmed by Connecticut Chemosensory Clinical Research Test (CCCRC-T).

Exclusion Criteria:

* Smokers
* Individuals with diagnosed rhinitis
* Individuals with diagnosed Neurological diseases
* Individuals submitted to brain surgery
* Previous historic of hyposmia and/ or anosmia
* Pregnancy
* Allergy to any of the substances present in the olfactory test kit
* Individuals who are undergoing another treatment for olfactory dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
To Assess the effectiveness of olfactory training therapy in the treatment of persistent olfactory dysfunctions after COVID-19 | 4 years
  The individuals of Experimental group 1 will be submitted to a olfactory training with essence oils, the participants will be reassessed with Olfactory test CCCRT monthly and this results will be compared with the reassessment results of the Experimental group 2 (no intervention group). The results of CCCRT of these two groups will be compared with Control group. The CCCRT olfactory test consists of n-butanol smell threshold test and smell identification test. Olfactory function score will be assessed (0: worst score; 7: best score).

SECONDARY OUTCOMES:
To Investigate by means of skull nuclear magnetic resonance (MRI) exams for possible neural correlates of olfactory dysfunctions present in post-COVID-19 patients | 4 years
  MRI imaging of olfactory bulb will be assessed in the individuals of this study, for better understanding of possible lesions at neural sites
To Measure by means of a standardized olfactory test the olfactory dysfunctions present in post-COVID-19 patients | 4 years
  CCCRT will be used to classify individuals as having normosmia, hyposmia or anosmia
Propose an olfactory training protocol appropriate to the demands of patients with post-COVID-19 olfactory dysfunction and in accordance with the reality of Brazilian public health services | 4 years
  The olfactory training using essence oils will be tested in this study as a low cost alternative for therapeutics

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade de Ensino E Assistência Em Fisioterapia E Terapia Ocupacional, Belém, Pará, Brazil